CLINICAL TRIAL: NCT03844191
Title: A Randomized Phase 1 Dose-Escalation Study in Healthy Volunteers and Subjects on Aspirin With Stable Coronary Artery Disease to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous RUC-4
Brief Title: A Randomized Phase 1 Dose-Escalation Study of Subcutaneously(SC) Administered RUC-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CeleCor Therapeutics (Industry)
Collaborators: Precision For Medicine (Industry); CirQuest Labs (Unknown); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEL-01
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — RUC-4 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The first 2 subjects in each dose cohort receive RUC-4 in a single- blind manner (only the subjects will blinded to treatment assignment), prior to randomizing the remaining 5 subjects to either RUC 4 (n = 4) or placebo (n = 1) in a double-blind manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Cohort 1 (Experimental): Cohort 1: 0.05 mg/kg RUC-4/placebo 7 subjects will be enrolled: 6 subjects will receive a single subcutaneous dose of RUC-4 and 1 subject will receive matched placebo.
  Interventions: Drug: RUC-4 Compound
- Part 1 Cohort 2 (Experimental): Cohort 2: 0.075 mg/kg RUC-4/placebo 7 subjects will be enrolled: 6 subjects will receive a single subcutaneous dose of RUC-4 and 1 subject will receive matched placebo.
  Interventions: Drug: RUC-4 Compound
- Part 2 Cohort 1 (Experimental): Cohort 1: initial dose to be selected by the Safety Review Committee (SRC) after completion of Part 1 (the same initial dose used in Part 1 or one of the previously studied higher doses that is lower than the overall RUC-4 BED) 7 subjects will be enrolled: 6 subjects will receive a single subcutaneous dose of RUC-4 and 1 subject will receive matched placebo.
  Interventions: Drug: RUC-4 Compound
- Part 2 Cohorts 2-3 (Experimental): 7 subjects (6 receiving RUC-4, 1 receiving placebo) will be enrolled in each dose cohort, with a safety evaluation performed after 2 subjects in a dose cohort receive RUC 4 and at the completion of dosing for all subjects in the dose cohort. Dose escalation to be determined by the SRC charter and will continue until identification of the overall RUC-4 BED or MTD
  Interventions: Drug: RUC-4 Compound
- Part 2 Dose Expansion Cohort 1 (Experimental): 14 subjects will receive a selected dose of RUC-4 based on SRC review of dose escalation data.
  In the expansion cohort, 7 subjects weighing 55 to 65 kg and 7 subjects weighing 100 to 120 kg will be enrolled; 12 subjects will receive a single subcutaneous dose of RUC-4 and 2 will receive matched placebo
  Interventions: Drug: RUC-4 Compound

INTERVENTIONS:
Drug: RUC-4 Compound — single subcutaneous administration of RUC-4
  Other Names: Placebo

SUMMARY:
This study is designed to assess tolerability of the weight-adjusted dose of RUC-4 (mg/kg) required to achieve 80% or more inhibition of the initial slope of platelet aggregation to 20 µM ADP by Light Transmission Aggregometry (LTA) within 15 minutes of SC administration of RUC-4 with return toward baseline values within 4 hours in healthy volunteers and subjects on aspirin with stable coronary artery disease (CAD). In the Dose Expansion Part, VerifyNow PRUTest will be used to measure platelet aggregation in addition to LTA.

Since the goal of RUC-4 therapy is to achieve maximal antiplatelet therapy as rapidly as possible, first the tolerability of the weight-adjusted dose (mg/kg) that inhibits ADP-induced platelet aggregation by 80% or more in 5 of 6 healthy volunteers will be identified. A similar dose escalation will be subsequently performed in subjects with CAD who are taking aspirin. To facilitate administration using a single weight-adjusted (mg/kg) dose for a defined group of subjects weighing between 55 and 120 kg, the study will also evaluate the safety and biologic effect on platelet aggregation of the weight adjusted (mg/kg) dose when administered to subjects with weights at either end of this range.

DETAILED DESCRIPTION:
Part 1 Dose Escalation:

Drug: RUC-4 0.05 mg/kg (Cohort 1) Drug: RUC-4 0.075 mg/kg (Cohort 2) Drug: Placebo (Cohorts 1-2)

Part 2 Dose Escalation Drug: RUC-4 (Cohort 1-3 doses to be defined) Placebo (Cohorts 1-3)

Part 2 Dose Expansion Drug: RUC-4 (dose to be defined, 1 Cohort) Drug: Placebo (1Cohort)

ELIGIBILITY:
Main Inclusion Criteria (all subjects)

* weight between 55-120 kg, inclusive, and BMI between 18-38 kg/m2
* females must be non-pregnant, non-lactating, and of non-childbearing potential.
* good general health as determined by no acute illness and no clinically significant abnormal findings on medical history, clinical laboratory test results, vital signs, or physical examination
* platelet count of 150,000/uL to 400,000/uL and mean platelet volume (MPV) within the normal range

Subjects with stable CAD, defined as history of documented myocardial infarction (MI) or angina, or evidence of CAD derived from cardiac stress test, or imaging (calcium score [greater than 100 or abnormal for age], angiography, computerized tomography, or magnetic resonance image); absence of angina, or presence of angina with no change in frequency, duration, precipitating causes or ease of relief for at least 60 days, and no ECG or biomarker evidence of myocardial damage in past 60 days

* blood pressure control achieved with 4 or fewer anti-hypertensive medications
* on a stable regimen of aspirin at a dose of 81 to 325 mg/day

Main exclusion criteria (all subjects):

* history of prior stroke or clinically significant cardiovascular (e.g., unstable angina, New York Heart Association [NYHA] class II, II or IV heart failure), dermatologic, endocrine, gastrointestinal (GI), hematologic, infectious, metabolic, neurologic, psychologic, or pulmonary disorder or any other condition, including active cancer that in the opinion of the PI would jeopardize the safety of the subject or impact the validity of the study results
* history of upper or lower GI bleeding requiring intervention or treatment within 12 months of Screening or endoscopic evidence of active peptic ulcer disease within 6 months of Screening
* bleeding score > 3 on the International Society on Thrombosis and Haemostasis Bleeding Assessment Tool
* coagulation abnormality, bleeding disorder, or history of documented prior hemorrhagic or thrombotic stroke
* whole blood donation and/or diagnostic blood evaluation exceeding 500 mL within 8 weeks of Screening
* surgical procedure, major injury, or dental procedure with high risk of bleeding within 30 days of Screening
* alcohol consumption of >210 mL of alcohol per week within 6 months of Screening, or alcohol detected in urine at Screening
* marijuana use within the past 3 months, or history/presence of substance abuse
* febrile illness within 14 days of Screening
* use of metformin within 7 days of Screening
* use of herbal or nutritional supplements/medicines within 7 days of Screening
* participation in another investigational product or device study within 30 days of Screening or during the study
* Presence of HIV antibody, HCV antibody, or HbsAg in serum at Screening
* employee of the Sponsor or The Lindner Center staff member directly affiliated with the study, or their immediate family member defined as spouse, parent, child, or sibling
* abnormal platelet aggregation or in vitro inhibition of platelet aggregation pattern by RUC-4
* receiving or have received in the past 30 days an anticoagulant or fibrinolytic agent
* a cardiac pacemaker
* history of allergy to any of the ingredients in the RUC-4 or placebo formulation

Healthy Subjects only:

* medication known to have an impact on platelet function within 30 days of Screening.
* abnormally low response to arachidonic acid-induced platelet aggregation
* screening ECG abnormality that is interpreted by the PI to be clinically significant

Stable CAD subjects only:

* medication known to have an impact on platelet function, with the exception of aspirin, within 30 days of Screening.

  ->4 anti-hypertensive medications required to achieve blood pressure control
* incomplete inhibition of arachidonic acid-induced platelet aggregation
* acute changes on ECG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Platelet Inhibition | 5 minutes
  inhibition of platelet aggregation
Platelet inhibition | 15 min
  inhibition of platelet aggregation
Platelet inhibition | 30 min
  inhibition of platelet aggregation
Platelet inhibition | 60 min
  inhibition of platelet aggregation
Platelet inhibition | 90 min
  inhibition of platelet aggregation
Platelet inhibition | 120 min
  inhibition of platelet aggregation
Platelet inhibition | 189 min
  inhibition of platelet aggregation
Platelet inhibition | 240 min
  inhibition of platelet aggregation
Platelet Inhibition | 360 min
  inhibition of platelet aggregation
Platelet Inhibition | 24 hours
  inhibition of platelet aggregation

CONTACTS AND LOCATIONS:
Locations (1):
- The Lindner Research Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kereiakes DJ, Henry TD, DeMaria AN, Bentur O, Carlson M, Seng Yue C, Martin LH, Midkiff J, Mueller M, Meek T, Garza D, Gibson CM, Coller BS. First Human Use of RUC-4: A Nonactivating Second-Generation Small-Molecule Platelet Glycoprotein IIb/IIIa (Integrin alphaIIbbeta3) Inhibitor Designed for Subcutaneous Point-of-Care Treatment of ST-Segment-Elevation Myocardial Infarction. J Am Heart Assoc. 2020 Sep;9(17):e016552. doi: 10.1161/JAHA.120.016552. Epub 2020 Aug 26. PMID 32844723